CLINICAL TRIAL: NCT04045990
Title: Neuromodulation of Language and Memory Networks in Alzheimer's Disease
Brief Title: Network Modulation in Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mark Eldaief, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2018P001362
Record Dates: First submitted 2018-08-29; First posted 2019-08-06 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Alzheimer Disease; Primary Progressive Aphasia; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Aphasia, Primary Progressive; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Patients with each condition will each undergo, in a crossover, within-subject design, two clocks of rTMS: active and SHAM.The order of active and SHAM blocks will be counterbalanced across subjects.
Who Masked: Participant
Masking Description: All participants will undergo SHAM stimulation as a control condition. They will be blinded as to whether they are receiving active or SHAM stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active stimulation (Experimental): Active rTMS will be administered with a MagPro X100 stimulator (MagVenture, Denmark), using a 70 mm figure-of-eight liquid cooled coil capable of doing active or sham stimulation (e.g. the Cool B70 coil or the Cool B65 A/P coil). Active rTMS will be delivered at 80-120% of a patient's resting or active motor threshold. rTMS will be administered in an excitatory pattern as 20Hz. Stimulation parameters will remain well within established safety guidelines (Rossi et al. 2009).
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- SHAM stimulation (Sham Comparator): SHAM stimulation will also be administered with a MagPro X100 stimulator (MagVenture, Denmark), using a 70 mm figure-of-eight liquid cooled coil capable of doing active or sham stimulation (e.g. the Cool B70 coil or the Cool B65 A/P coil). SHAM rTMS will be delivered at 80-120% of a patient's resting or active motor threshold. SHAM stimulation will be delivered to the exact same cortical targets as active rTMS. While no electromagnetic stimulation will be delivered during SHAM, the sounds will approximate active stimulation and skin electrodes will approximate the sensation of active rTMS. Inclusion of a sham condition in this protocol is critical to measure whether or not the stimulation is improving memory or language performance, or whether practice effects or other non-specific effects are responsible for any changes in memory or language performance which may be observed.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — rTMS is a method to focally and reversibly stimulate a pre-specified cortical target. rTMS works through the principle of electromagnetic induction.

SUMMARY:
The purpose of this study is to assess the effects of non-invasive brain stimulation on memory and language ability in patients with two phenotypic variations of underlying Alzheimer disease pathology: amnestic mild cognitive impairment (aMCI) and logopenic variant of primary progressive aphasia (lvPPA). This study will use repetitive Transcranial Magnetic Stimulation (rTMS) to stimulate nodes of networks that are thought to be affected in these two conditions. Specifically, a node of the Default Mode Network (DMN)-the angular gyrus (AG)-will be stimulated in aMCI patients; and a node of the language network-the posterior inferior frontal gyrus (pIFG) will be stimulated in patients with lvPPA.

We will use functional connectivity MRI (fcMRI) to assess changes in functional network architecture following the stimulation. We will also assess putative cognitive improvements resulting from the stimulation by in-depth language testing in lvPPA patients and in-depth memory testing in aMCI patients.

DETAILED DESCRIPTION:
Specific Aims

Aim 1: To investigate the feasibility of selective rTMS modulation of the Default Mode Network (DMN) vs. language network in patients with aMCI and lvPPA. We will assess the reliability of the rTMS/fcMRI approach to network modulation by studying the same subjects over repeated sessions, with the same methodology, including appropriate sham stimulation conditions.

Hypothesis 1a: Changes in network functional connectivity following excitatory rTMS to AG (a node of the DMN) and pIFG (a node of the language network) across identical stimulation sessions separated in time, will show minimal within subject variability in aMCI and lvPPA patients, respectively, thus confirming the reliability of the approach and the reproducibility of prior findings demonstrating connectivity changes within the DMN and language networks.

Hypothesis 1b: High frequency rTMS to pIFG will reliably increase pIFG-SMG-pMTG functional connectivity within the language network; high frequency rTMS to AG will reliably increase functional connectivity between pIPL and HF in the DMN.

Hypothesis 1c: The changes in network functional connectivity will be selective, in that stimulation to AG (in the DMN) will not modulate connectivity within the language network, while stimulation to pIFG (in the language network) will not modulate DMN connectivity.

Aim 2: To assess the effects of rTMS modulation on memory and language function in patients with aMCI and lvPPA.

Hypothesis 2a: Excitatory rTMS to the language network will be associated with improved language performance in patients with lvPPA.

Hypothesis 2b: Excitatory rTMS to the DMN will be associated with improved memory performance in patients with aMCI.

Hypothesis 2c: Cognitive improvements will persist for at least two weeks following cessation of rTMS.

Aim 3: To identify the functional network mechanisms underlying cognitive improvement in patients with aMCI and lvPPA after rTMS.

Hypothesis 3a: Alterations in intrinsic functional connectivity (as assessed with fcMRI) within each network following rTMS will correlate with improved cognitive performance.

Hypothesis 3b: Patients with a greater degree of atrophy and tau pathology within each network (assessed in a prior study) at baseline will predict a lesser response to rTMS.

We will recruit up to 20 patients with aMCI and up to 20 patients with lvPPA (with amyloid and tau imaging or CSF biomarkers supportive of underlying AD pathology). We will first perform a baseline functional connectivity MRI (fcMRI), the purpose of which will be to obtain individualized network maps which can be used to target the networks of interest during future sessions.

This will be followed by up to two weeks of five consecutive days of stimulation (Monday through Friday). aMCI patients will receive stimulation to the angular gyrus (AG) node of the DMN, and lvPPA patients will receive stimulation to the posterior inferior frontal gyrus (pIFG) node of the language network. During one of the two weeks stimulation will be active, and during the other week stimulation will be SHAM. Order of active and SHAM stimulation blocks will be counterbalanced.

We will concomitantly assess the effects of rTMS modulation on memory and language function in patients with aMCI and lvPPA, and in so doing identify the functional network mechanisms underlying cognitive improvement after rTMS. Language and memory assessments will be performed on days 1 (Monday) , 3 (Wednesday) and 5 (Friday) of the week. Finally, to assess the distributed effects of the stimulation upon functional connectivity, fcMRI will be performed on days 1 (Monday) and 5 (Friday).

We anticipate these results will lead to an impactful manuscript showing proof-of-concept data: 1) that it is possible to improve memory in aMCI and language in lvPPA using rTMS targeted selectively to the relevant brain network, and: 2) regarding mechanisms underlying the effects of rTMS on network function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, age 18-90, who carry a diagnosis of either the logopenic variant (lvPPA) of PPA or amnestic MCI (aMCI). Patients must have been observed for at least one year by a specialized clinician.
2. The presence of underlying AD pathology must be verified by a prior amyloid-PET and/or Tau-PET imaging (done as part of a prior protocol), or CSF biomarkers of AD pathology.
3. Patients with lvPPA must have at least mild to moderate language impairment.
4. Patients with aMCI must meet criteria for this condition, including the presence of at least mild to moderate episodic memory impairment.
5. Patients must be native English speakers.
6. Patients must have a study partner (e.g. spouse, sibling, adult child, friend) who can accompany them to all study visits.

Exclusion Criteria:

1. Any history of seizures, unexplained loss of consciousness or a first-degree family member with epilepsy (to ensure safety to receive rTMS).
2. Any history of significant co-occurring neurological illness unrelated to the neurodegenerative disease in question (e.g. multiple sclerosis), or significant medical problems (e.g. poorly controlled diabetes/hypertension or cancer within 5 years).
3. Active symptoms of major depressive disorder, bipolar disorder, schizophrenia, substance use disorder or significant premorbid intellectual disability according to DSM criteria.
4. MRI evidence of significant (e.g. confluent leukoariosis or stroke) cerebrovascular disease, hydrocephalus or the presence of a space-occupying intra-cranial mass.
5. Contraindications to MRI or rTMS including: cardiac pacemaker or pacemaker wires, neurostimulators, implanted pumps, metal in the body (rods, plates, screws, shrapnel, dentures, IUD), surgical aneurysm clips in the head, previous neurosurgery or cochlear implants.
6. In line with published MGH IRB guidelines for rTMS, pregnancy must be ruled out by urine ß-HCG if answers to screening questions suggest that pregnancy is possible and if female participants are premenopausal and of child-bearing age. Subjects will not be able to enroll if they are breastfeeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Boston Naming Test | Up to 5 weeks
  A test of confrontation naming of drawn pictures.
Western Aphasia Battery-repetition | Up to 5 weeks
  A test of the ability to repeat phonetically complex phrases
Western Aphasia Battery-reading comprehension | Up to 5 weeks
  A test of the ability to correctly comprehend read material
Western Aphasia Battery-spelling | Up to 5 weeks
  A test of the ability to spell irregular words.
Controlled Oral Word Association Test | Up to 5 weeks
  A test of word generation, e.g. generation of as many words as possible beginning with a certain letter of the alphabet.
Cambridge Semantic Battery | Up to 5 weeks
  A test of semantic knowledge through word-pairings.
The Northwestern Anagram Test | Up to 5 weeks
  A test of non-verbal production of sentences.
Picture Description Test | Up to 5 weeks
  A test in which patients write a paragraph describing a picture, such as a picnic or the cookie theft picture.
Changes in intrinsic functional connectivity | Up to 5 weeks
  Changes in region-to-region functional connectivity within the stimulated networks will be assessed, e.g. changes in connectivity in the DMN will be assessed in aMCI patients and changes in the language network will be assessed in lvPPA patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with researchers outside of this protocol.